CLINICAL TRIAL: NCT00786630
Title: Intervention to Reduce Injection Drug Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-1131; 2R01DA009832-11 (NIH)
Record Dates: First submitted 2008-11-04; First posted 2008-11-06 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Substance Abuse
Keywords: Drug treatment entry and retention; Drug injection frequency; HIV risk behaviors; Hepatitis C risk behaviors
MeSH Terms: conditions — Substance-Related Disorders | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case Management (Experimental)
  Interventions: Behavioral: Strengths-based case management
- Facilitated Treatment Alliance (Experimental)
  Interventions: Behavioral: Case management plus facilitated treatment alliance

INTERVENTIONS:
Behavioral: Strengths-based case management — Clients will receive counseling and/or referrals for help with nine life domains (life skills, finances, leisure activities, relationships, living arrangements, occupation/education, health, mental health, recovery from substances, legal assistance) for a period of five months after baseline.
  Arms: Case Management
Behavioral: Case management plus facilitated treatment alliance — Clients will receive counseling and/or referrals for help with nine life domains (life skills, finances, leisure activities, relationships, living arrangements, occupation/education, health, mental health, recovery from substances, legal assistance) for a period of five months after baseline. They will also receive a facilitated treatment alliance, which consists of meetings with methadone counselors to aid in treatment entry.
  Arms: Facilitated Treatment Alliance

SUMMARY:
This is a five-year prospective randomized trial comparing two intervention conditions designed to facilitate substance abuse treatment entry and enhance retention in order to reduce the behaviors associated with HIV and HCV risk among injection drug users (IDUs) and to improve client overall functioning. The overall goal of this project is to compare strengths-based case-management (CM) to an enhanced version of CM that uses case managers to facilitate a therapeutic alliance (CM/FTA) among out-of-treatment IDUs in Denver.

ELIGIBILITY:
Inclusion Criteria:

* opiate injection at least 3 times a week during the last 6-months
* 18 years of age or older
* no drug abuse treatment in the 30-days prior to the interview
* not transient
* no known reason (e.g. pending jail time) why they will not be available for follow-up interviews
* not involved in Project Safe research activities in the previous 12 months
* willing to meet with an Addiction Research and Treatment Services (methadone clinic) counselor
* eligible to be treated at ARTS

Exclusion Criteria:

* too intoxicated or impaired mentally to voluntarily consent to participate in the project and/or respond to the interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 726 (Actual)
Dates: Start 2007-11; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Treatment entry and retention | Baseline, 6 months after baseline, 12 months after baseline

SECONDARY OUTCOMES:
Drug injection and HIV/HCV risk behaviors | Baseline, 6 months after baseline, 12 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Robert E. Booth, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- Project Safe, Denver, Colorado, United States